CLINICAL TRIAL: NCT00149058
Title: A Phase II Randomised Trial to Investigate the Safety and Efficacy of Recombinant Human Erythropoietin on Infarct Size in Patients Undergoing Primary Percutaneous Coronary Angioplasty for ST-Segment Elevation Myocardial Infarction
Brief Title: Erythropoietin in Acute Myocardial Infarction
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hammersmith Hospitals NHS Trust (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 05/MREC00/7
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2005-09-08 (Estimated); Status verified 2005-09

CONDITIONS: Acute Myocardial Infarction
Keywords: acute myocardial infarction; primary angioplasty
MeSH Terms: interventions — Erythropoietin

INTERVENTIONS:
Drug: Erythropoietin

SUMMARY:
Erythropoietin (EPO) is a naturally occuring hormone which regulates the body's response to lack of oxygen and controls the number of red cells in the blood. Recent studies in animals have shown that EPO has protective effects when organs such as the heart and brain are injured by lack of oxygen due to reduced blood supply.

We wish to test the idea that giving a patient, who is having a heart attack, an injection of EPO will reduce the size of the heart attack.

DETAILED DESCRIPTION:
We wish to perform a randomised double-blind, placebo-controlled clinical trial to examine the effects of EPO given at the time of primary angioplasty for acute myocardial infarction (MI) on myocardial infarct size. In this trial the null hypothesis is that there is no effect of EPO on myocardial infarct size, the alternative hypothesis is that EPO reduces myocardial infarct size.

124 subjects with acute ST-elevation MI who fulfil the inclusion/exclusion criteria and give informed consent to participate in the study will be recruited from patients referred to the cardiac catheterisation laboratories at the Hammersmith Hospital and King's College Hospital. Subjects will undergo primary percutaneous coronary angioplasty (primary PCI) according to standard clinical protocols. Subjects will be randomised to either placebo or EPO at the time of primary PCI. EPO will be given as a bolus of 12ml containing 33,000U over 30 mins via a peripheral vein followed by an infusion of 24ml containing 67,000 U over 12 hours. Placebo will be identical to EPO without the active ingredient. After the PCI subjects will receive standard care on the coronary care unit. An additional 20ml of blood will be taken each day at the time of routine clinical venesection for storage and subjects will have gadolinium enhanced cardiovascular magnetic resonance (CMR) performed before discharge to evaluate infarct size. Follow-up will be performed at 30 days (clinical, ECG and 20ml blood sample) and at 90 days (clinical, ECG and CMR scan and blood sample). The study will end at 90 days and patients will continue with standard clinical care under the direction of a consultant cardiologist.

CMR will be performed in the Robert Steiner MR Unit/Imaging Department, Hammersmith Hospital using a 1.5 tesla scanner according to standard protocols. Each scan will last about 1h and information will be collected on tissue characteristics, left ventricular function, wall motion abnormalities, myocardial perfusion. Myocardial infarcts will be detected by late contrast gadolinium enhancement. Gadolinium will be used at doses up to 0.2mmol/kg and is safe with an incidence of mild and transient side effects including headache and nausea of ~1%. Scans will be performed with under continuous ECG monitoring with a doctor and at least 1 other person present. Resuscitation facilities will be available at all times and the MRI facility is covered by an experienced 24 hour a day cardiac arrest team.

ELIGIBILITY:
Inclusion Criteria:

* Male or female >18 years of age
* Weight between 50 kg and 120 kg
* Suspected of having his/her first-documented STEMI
* Symptoms of ischemia of >20 min with < 6h prior to PCI
* Either 1mm ST elevation in at least two contiguous limb leads or >2mm ST elevation in 2 contiguous chest leads
* Primary PCI to occur within 8h from the onset of symptoms
* Women of childbearing potential must have a negative pregnancy test

Exclusion Criteria:

* Contraindications to MRI scanning
* History or ECG evidence of previous STEMI
* Cardiogenic shock
* NYHA class III-IV heart failure
* LBBB or AF on ECG; 6.Major trauma, major surgery, eye, spinal cord, or brain surgery within the last 3 months
* Significant hepatic disturbance
* Chronic renal impairment (Creatinine >200µmol/L)
* Stroke or TIA <6 months
* Pregnancy or breast-feeding
* Dependence on alcohol or other DOA
* Significant psychiatric/neurologic disease that would prevent adherence to the requirements of the protocol
* Significant immunocompromise (including, but not limited to AIDS and immune-suppressive therapy
* Current treatment with human recombinant erythropoietin
* Current hemodialysis or peritoneal dialysis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124
Dates: Start 2005-10; Study Completion 2008-01

PRIMARY OUTCOMES:
Myocardial infarct size

SECONDARY OUTCOMES:
Death
Reinfarction

CONTACTS AND LOCATIONS:
Overall Officials: Jaspal S Kooner, Principal Investigator — Hammersmith Hospitals NHS Trust
Locations (2):
- United Kingdom (2):
  - Hammersmith Hospital NHS Trust, London
  - King's College London, London